CLINICAL TRIAL: NCT03586427
Title: A Double-Blind, Placebo-Controlled, Fixed-Dose Study of AGN-241751 in Adult Participants With Major Depressive Disorder
Brief Title: AGN-241751 in the Treatment of Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Syndeio Biosciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3125-201-002
Record Dates: First submitted 2018-06-22; First posted 2018-07-13 (Actual); Results first posted 2022-08-02 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- AGN-241751 Dose 1 (Experimental): AGN-241751 Dose 1 administered as 1 tablet taken orally every day
  Interventions: Drug: AGN-241751
- AGN-241751 Dose 2 (Experimental): AGN-241751 Dose 2 administered as 1 tablet taken orally every day
  Interventions: Drug: AGN-241751
- AGN-241751 Dose 3 (Experimental): AGN-241751 Dose 3 administered as 1 tablet taken orally every day
  Interventions: Drug: AGN-241751
- AGN-241751 Dose 4 (Experimental): AGN-241751 Dose 4 administered as 1 tablet taken orally every day
  Interventions: Drug: AGN-241751
- Placebo (Placebo Comparator): Placebo administered as 1 tablet taken orally every day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AGN-241751 — AGN-241751 administered orally as a single tablet
  Arms: AGN-241751 Dose 1; AGN-241751 Dose 2; AGN-241751 Dose 3; AGN-241751 Dose 4
Drug: Placebo — Placebo administered orally as a single tablet
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy at 1 day post initial oral dose of AGN-241751 compared with placebo in participants with Major Depressive Disorder (MDD).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from the participant has been obtained prior to any study -related procedures (as described in Appendix 3).
* Male or female participants must be 18 to 65 years of age, inclusive, at the time of signing the informed consent.
* Meet Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria for MDD (based on confirmation from the modified Structured Clinical Interview for DSM disorders [SCID]), with a current major depressive episode of at least 8 weeks and not exceeding 18 months in duration at Visit 1.
* Have a minimum score of 26 on the rater-administered Montgomery-Asberg depression rating scale (MADRS) and a minimum score of 24 on the computer-administered MADRS at both Visit 1 (Screening) and Visit 2 (Baseline).
* Have a difference of no greater than 7 points between the rater-administered MADRS and computer-administered MADRS at both Visit 1 (Screening) and Visit 2 (Baseline).
* Have a clinical global impression-severity (CGI-S) score ≥ 4 at both Visit 1 (Screening) and Visit 2 (Baseline).
* Have a negative serum β-human chorionic gonadotropin (β-hCG) pregnancy test if a woman of childbearing potential (WOCBP).
* Female participants willing to minimize the risk of becoming pregnancy for the duration of the clinical study and follow-up period. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:
* not a WOCBP OR
* A WOCBP who agrees to follow the contraceptive guidance in Appendix 5 of protocol during the treatment period and for at least 5 terminal half-lives after the last dose of study treatment.
* Male participants willing to minimize the risk of inducing pregnancy for the duration of the clinical study and follow-up period. A male participant must agree to use contraception as detailed in Appendix 5 of this protocol during the treatment period and for at least 5 terminal half-lives after the last dose of study treatment and refrain from donating sperm during this period.
* Able, as assessed by the investigator, and willing to follow study instructions and likely to complete all required study visits.
* Normal physical-examination findings, clinical-laboratory test results, and electrocardiogram (ECG) results from Visit 1 (Screening) or abnormal results that are determined to be not clinically significant by the investigator.
* Body mass index (BMI) within the range 18 and 40 kg/m^2 (inclusive).
* Eligibility confirmed through a formal adjudication process (see Section 9 Diagnostic Assessments).

Exclusion Criteria:

Psychiatric and Treatment-Related Criteria

* DSM-5-based diagnosis of any disorder other than MDD that was the primary focus of treatment within 6 months before Visit 1. Comorbid generalized anxiety disorder, social anxiety disorder, or specific phobias are acceptable provided they play a secondary role in the balance of symptoms and are not the primary driver of treatment decisions.
* Lifetime history of meeting DSM-5 criteria for:
* Schizophrenia spectrum or other psychotic disorder
* Bipolar or related disorder
* Major neurocognitive disorder
* Neurodevelopmental disorder of greater than mild severity or of a severity that impacts the participant's ability to consent, follow study directions, or otherwise safely participate in the study
* Dissociative disorder
* Posttraumatic stress disorder
* MDD with psychotic features
* History of meeting DSM-5 criteria for alcohol or substance use disorder (other than nicotine or caffeine) within the 6 months before Visit 1.
* DSM-5-based diagnosis of any personality disorder of sufficient severity to interfere with participation in this study in the opinion of the investigator.
* History (based on participant report and/or medical records, and investigator judgment) of:
* Inadequate response to electroconvulsive therapy (ECT), a monoamine oxidase inhibitor, ketamine, or adjunctive treatment with an antipsychotic
* Treatment with clozapine or any depot antipsychotic
* ECT, vagus nerve stimulation, transcranial magnetic stimulation, or any experimental central nervous system treatment during the current episode or in the 6 months before Visit 1 (whichever is longer)
* Tardive dyskinesia, serotonin syndrome, or neuroleptic malignant syndrome
* Having received:
* Anticonvulsant/mood stabilizer, within 1 year prior to Visit 1
* Antipsychotic in the current episode, with the exception of quetiapine given for insomnia ≤ 50 mg/day provided it can be safely discontinued prior to Visit 2
* Combination therapy of 2 or more antidepressant therapies (ADTs) in the current episode if given for depression at adequate dose and duration
* ADT augmentation agent in the current episode
* Lifetime history of nonresponse to ≥ 2 antidepressants after adequate trials (adequate treatment is defined as at least 6 weeks at an adequate dose(s) based on approved package insert recommendations) or a non-response to an antidepressant after adequate treatment for the current major depressive episode.
* Positive result at Visit 1 from the urine drug screen (UDS) test for any prohibited medication. Exception: participants with a positive UDS at Visit 1 for opiates, cannabinoids, or episodic use of benzodiazepines may be allowed in the study provided:
* The drug was used for a legitimate medical purpose;
* The drug can be discontinued prior to participation in the study (except for episodic use of benzodiazepines which may be continued); and
* A repeat UDS is negative for these substances prior to enrollment (except for episodic use of benzodiazepines which may be continued)
* Suicide risk, as determined by meeting any of the following criteria:
* A suicide attempt within the past year
* Significant risk, as judged by the investigator, based on the psychiatric interview or information collected in the C-SSRS at Visit 1 (Screening) or Visit 2 (Baseline)
* MADRS Item 10 score ≥ 5 at Visit 1 (Screening) or Visit 2 (Baseline) on the MADRS
* At imminent risk of injuring self or others or causing significant damage to property, as judged by the investigator.
* Requiring concomitant treatment with any of the prohibited medications, supplements, or herbal products listed in Appendix 6 of protocol, including any psychotropic drug or any drug with psychotropic activity, except as described in Section 7.7.2. of protocol.
* Prior participation in any investigational study of AGN-241751.
* Initiation or termination of psychotherapy for depression within the 3 months preceding Visit 1, or plans to initiate, terminate, or change such therapy during the course of the study. (Support meetings or counselling [eg, marital counselling] are allowed provided they are no more frequent than weekly and do not have treatment of depression as their objective).
* Ongoing treatment with phototherapy, or termination of phototherapy within 1 month of Visit 1.
* Known allergy or sensitivity to the study medication or its components.

Other Medical Criteria

* BMI < 18 kg/m^2 or > 40 kg/m^2 at screening.
* Females who are pregnant, breastfeeding, or planning to become pregnant or breastfeed during the study.
* WOCBP and male partners of WOCBP, not using a reliable means of contraception (Appendix 5 of protocol).
* Participant has a condition or is in a situation which, in the investigator's opinion, may put the participant at significant risk, may confound the study results, or may interfere significantly with the participant's participation in the study.
* Any cardiovascular disease that is clinically significant, unstable, or decompensated.
* Heart rate (supine) of ≤ 45 beats per minute (bpm) or ≥ 120 bpm, or any heart rate that is clinically symptomatic at Visit 1 or Visit 2 based upon vital signs.
* Any systolic and/or diastolic blood pressure (BP) that is symptomatic or clinically significant in the opinion of the investigator.
* History of congenital QTc prolongation or QTc prolongation (screening ECG with QTcF ≥ 450 msec for men and QTcF ≥ 470 msec for women).
* Hypothyroidism or hyperthyroidism, unless stabilized on appropriate pharmacotherapy with no change in dosage for at least 1 month before Visit 1.
* History of seizure disorder, stroke, significant head injury, tumor of the central nervous system, or any other condition that predisposes to seizure.
* Known human immunodeficiency virus (HIV) infection.
* Positive hepatitis C antibody on screening, with the exception of participants for whom the reflex hepatitis C virus ribonucleic acid (HCV RNA) test is negative.
* Positive test for hepatitis B surface antigen and/or hepatitis B core antibody immunoglobulin M.
* Screening liver enzyme test (aspartate aminotransferase [AST] and/or alanine aminotransferase [ALT]) results > 2 times the upper limit of normal (ULN).

Other Criteria

* Current enrollment in an investigational drug or device study or participation in such a study within 6 months of entry into this study.
* Employee, or immediate relative of an employee, of the sponsor, any of its affiliates or partners, or the study center.
* Inability to speak, read, and understand the English language sufficiently to understand the nature of the study, to provide written informed consent, or to allow the completion of all study assessments.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2018-06-13 (Actual); Primary Completion 2019-07-22 (Actual); Study Completion 2019-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald M Burch, MD PhD, Study Director — Syndeio Biosciences, Inc
Locations (25):
- United States (25):
  - Health Initiatives Research PLLC, Fayetteville, Arkansas
  - Synexus US - Cerritos, Cerritos, California
  - Wake Research - Pharmacology Research Institute, Encino, California
  - Wake Research - Pharmacology Research Institute, Newport Beach, California
  - Pacific Research Partners, LLC, Oakland, California
  - North County Clinical Research, Inc., Oceanside, California
  - Collaborative Neuroscience Network, Torrance, California
  - Elite Clinical Trials, Inc., Wildomar, California
  - Synexus US - Atlanta, Atlanta, Georgia
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Pillar Clinical Research, Lincolnwood, Illinois
  - Boston Clinical Trials, Boston, Massachusetts
  - Hassman Research Institute, Berlin, New Jersey
  - Center for Emotional Fitness, Cherry Hill, New Jersey
  - Neurobehavioral Research, Inc, Cedarhurst, New York
  - Synexus US - Queens, Jamaica, New York
  - Eastside Comprehensive Medical Center, New York, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Neuro-Behavioral Clinical Research, Inc, North Canton, Ohio
  - IPS Research, Oklahoma City, Oklahoma
  - Clinical Neuroscience Solutions, Inc - Memphis, TN, Memphis, Tennessee
  - Research Strategies of Memphis, LLC, Memphis, Tennessee
  - Donald J. Garcia, Jr., MD, PA, Austin, Texas
  - FutureSearch Trials of Dallas, LP, Dallas, Texas
  - Northwest Clinical Research Center, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: No
This is a phase 2 dose finding proof of concept study therefore data will not be shared.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After providing written consent, participants entered a single-blind placebo lead-in screening period of up to 7 days. Participants received single-blind placebo during the screening period. Participants meeting the eligibility criteria at the end of the screening period were randomized into one of the 5 treatment groups and entered the double-blind treatment period.
Groups:
- AGN-241751 Dose 1: AGN-241751 Dose Level 1: 0.25 mg weekly for 3 weeks
- AGN-241751 Dose 2: AGN-241751 Dose Level 2: 1 mg weekly for 3 weeks
- AGN-241751 Dose 3: AGN-241751 Dose Level 3: 3 mg weekly for 3 weeks
- AGN-241751 Dose 4: AGN-241751 Dose Level 4: 10 mg weekly for 3 weeks
- Placebo: Placebo: Placebo administered weekly as a single tablet and daily to all groups except for drug day one time each week
Period: Overall Study
Arm/Group | AGN-241751 Dose 1 | AGN-241751 Dose 2 | AGN-241751 Dose 3 | AGN-241751 Dose 4 | Placebo
Started | 48 | 50 | 52 | 50 | 51
Completed | 48 | 46 | 46 | 46 | 46
Not Completed | 0 | 4 | 6 | 4 | 5
Not completed — Lost to Follow-up | 0 | 3 | 1 | 3 | 3
Not completed — Withdrawal by Subject | 0 | 1 | 2 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 1
Not completed — Noncompliance with study drug | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- AGN-241751 Dose 1: AGN-241751 0.25 mg administered as 1 tablet taken orally one time each week for 3 weeks
  Placebo administered as 1 tablet taken orally every day except days AGN-214751 was taken
- AGN-241751 Dose 2: AGN-241751 1 mg administered as 1 tablet taken orally one time each week for 3 weeks
  Placebo administered as 1 tablet taken orally every day except days AGN-214751 was taken
- AGN-241751 Dose 3: AGN-241751 3 mg administered as 1 tablet taken orally one time each week for 3 weeks
  Placebo administered as 1 tablet taken orally every day except days AGN-214751 was taken
- AGN-241751 Dose 4: AGN-241751 10 mg administered as 1 tablet taken orally one time each week for 3 weeks
  Placebo administered as 1 tablet taken orally every day except days AGN-214751 was taken
- Total: Total of all reporting groups
Arm/Group | AGN-241751 Dose 1 | AGN-241751 Dose 2 | AGN-241751 Dose 3 | AGN-241751 Dose 4 | Placebo | Total
Number analyzed (Participants) | 48 | 50 | 52 | 50 | 51 | 251
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.8 (14.02) | 41.8 (13.53) | 42.2 (14.23) | 42.9 (13.48) | 40.0 (14.49) | 41.7 (13.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 15 | 16 | 20 | 30 | 114
  Male | 15 | 35 | 36 | 30 | 21 | 137
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 1
  Asian | 3 | 1 | 1 | 2 | 1 | 8
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 1
  Black or African American | 18 | 24 | 22 | 15 | 20 | 99
  White | 24 | 24 | 28 | 32 | 27 | 135
  More than one race | 1 | 1 | 1 | 0 | 2 | 5
  Unknown or Not Reported | 1 | 0 | 0 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 48 | 50 | 52 | 50 | 51 | 251
Current antidepressant usage [Count of Participants; unit: Participants] | 7 | 13 | 13 | 13 | 11 | 57

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score
Description: The MADRS is a clinician-rated scale to assess depressive symptomatology during the preceding week. Participants are rated on 10 items (feelings of sadness, lassitude, pessimism, inner tension, suicidality, reduced sleep or appetite, difficulty concentrating, and lack of interest) each on a 7-point scale from 0 (no symptoms) to 6 (symptoms of maximum severity). The total score ranges from 0 to 60 with a higher score indicating more depression. A negative change score indicates improvement.
Time Frame: Baseline to Day 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | AGN-241751 Dose 1 | AGN-241751 Dose 2 | AGN-241751 Dose 3 | AGN-241751 Dose 4 | Placebo
Number analyzed (Participants) | 48 | 50 | 52 | 50 | 51
score on a scale | -8.6 (1.21) | -8.0 (1.19) | -9.5 (1.18) | -10.6 (1.18) | -7.7 (1.18)
Statistical Analysis 1: Comparison: AGN-241751 Dose 1 vs AGN-241751 Dose 2 vs AGN-241751 Dose 3 vs AGN-241751 Dose 4 vs Placebo; Each dose group was compared to placebo; Test type: Other — Mixed model of repeated measures least square estimates of change compared to placebo; p > 0.05, Mixed Models Analysis — Comparison of each dose level change from baseline to placebo baseline yielded P values >0.05

2. Secondary Outcome: Change From Baseline in MADRS Total Score at Week 3
Description: as for outcome 1
Time Frame: Baseline to Week 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | AGN-241751 Dose 1 | AGN-241751 Dose 2 | AGN-241751 Dose 3 | AGN-241751 Dose 4 | Placebo
Number analyzed (Participants) | 48 | 50 | 52 | 50 | 51
score on a scale | -11.5 (1.56) | -12.5 (1.54) | -14.1 (1.55) | -13.5 (1.54) | -13.6 (1.54)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | AGN-241751 Dose 1 | AGN-241751 Dose 2 | AGN-241751 Dose 3 | AGN-241751 Dose 4 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/50 | 0/52 | 0/50 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/50 | 0/52 | 0/50 | 0/51
Other Adverse Events (participants affected / at risk) | 17/48 | 18/50 | 12/52 | 19/50 | 16/51
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AGN-241751 Dose 1 (N=48) | AGN-241751 Dose 2 (N=50) | AGN-241751 Dose 3 (N=52) | AGN-241751 Dose 4 (N=50) | Placebo (N=51)
Headache (Nervous system disorders) | 3 (3) | 3 (3) | 3 (3) | 2 (2) | 4 (4)
Somnolence (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 3 (3) | 3 (3) | 2 (2)
Sedation (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (2) | 1 (1) | 2 (2)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Insomnia (Nervous system disorders) | 0 (0) | 5 (5) | 0 (0) | 1 (1) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral Upper Respiratory Infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-05-01): https://cdn.clinicaltrials.gov/large-docs/27/NCT03586427/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-03): https://cdn.clinicaltrials.gov/large-docs/27/NCT03586427/SAP_001.pdf